CLINICAL TRIAL: NCT05248503
Title: Impact of Complex Care Training of Hereditary Epidermolysis Bullosa on Caregiver Burden (FIREB)
Acronym: FIREB
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211522
Record Dates: First submitted 2022-01-17; First posted 2022-02-21 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Hereditary Epidermolysis Bullosa
Keywords: hereditary epidermolysis bullosa; nursing care; care training; child

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Nurse: Pediatric nurses taking charge of the care of patients with epidermolysis bullosa at Necker Hospital
  Interventions: Behavioral: Complex Care Training of Hereditary Epidermolysis Bullosa

INTERVENTIONS:
Behavioral: Complex Care Training of Hereditary Epidermolysis Bullosa — Training in the care of epidermolysis bullosa by combining theoretical content on the disease and practical workshops.

SUMMARY:
Hereditary epidermolysis bullosa (EBH) is a rare, orphan disease characterized by skin and mucous membrane fragility.

The latest scientific data show that the proposed treatments are still in the experimental stage and that no curative treatment is available. The repercussions of this chronic disease, with neonatal onset, are major.

Epidermolysis bullosa requires multidisciplinary medical management, nursing care, psychological and social care.

Skin care involves preventing and treating chronic wounds and identifying their complications. The very great cutaneous-mucous fragility makes these treatments painful, long and complex, the caring hand itself being able to cause new wounds. Analgesics of different levels are not effective enough during treatment.

Along with counseling and education, nursing takes a central role in multi-professional accompaniment interventions to support and relieve families.

Parents became home caregivers out of necessity, and developed specific skills in epidermolysis bullosa, their child and dressings. They have great and demanding expectations of caregivers facing this rare disease, for which they are not trained in their degree course. Despite the severe nature of the disease, few studies have been carried out on the impact and psychosocial consequences on patients and their families, yet there is an expressed need for support.

The burden on parents is heavy, assessed by specific scales, but to date there are no studies examining the impact of epidermolysis bullosa care on caregiver stress.

ELIGIBILITY:
Inclusion Criteria:

* Nurse, nursing assistant, nursery nurse, childcare assistant, state graduates caring for patients with EBH and working at Necker Hospital.
* Having participated in the entire training program specific to the complex care of epidermolysis bullosa.
* Informed and not opposed to their participation in research.

Exclusion Criteria

* Person under tutorship or curatorship.
* Other health professionals (physiotherapist, doctor, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any caregiver who, within their department, must take charge of the complex care of patients with EBH (nurse, caregiver, pediatric nurse, childcare assistant) is eligible.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change of anxiety level | Change form baseline (before training) and at the end of the second day of training
  Anxiety will be assessed using the Anxiety - Spielberger State self-quiz, rated from 20 to 80 (80 indicating maximum anxiety state).

SECONDARY OUTCOMES:
Anxiety evolution | 3 months after training
  Anxiety will be assessed using the Anxiety - Spielberger State self-quiz, rated from 20 to 80 (80 indicating maximum anxiety state).
Anxiety auto-evaluation | Before training. 3 and 6 months after the training
  Self-assessment of factors that may induce anxiety measured on a Likert Scale from 0 to 4 (4 indicating a factors induces an high level of anxiety)
Feeling of skills | Before training. 3 and 6 months after the training
  Self-assessment of feeling of skills on Likert scales from 0 to 4 (4 indicating a factors induces an high level of anxiety)
Nurse knowledge about Epidermolysis bullosa | Before and after the training. 3 and 6 months after the training
  A true/false questionnaire with degree of certainty assessing knowledge about epidermolysis bullosa
Satisfaction questionnaire | At the end of the second day of training.
  Satisfaction questionnaire on the quality and content of the training with a Likert scale ( 0 to 5; an higher score indicates better outcome) and open questions.

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine COMPAIN, RN, Principal Investigator — Necker Hospital, APHP
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ingen-Housz-Oro S, Blanchet-Bardon C. Épidermolyses bulleuses héréditaires. EMC - Dermatol-Cosmétologie. 1 févr 2004 ; 1(1) :2 18.
- [Background] Chiaverini C, Bourrat E, Mazereeuw-Hautier J, Hadj-Rabia S, Bodemer C, Lacour JP. [Hereditary epidermolysis bullosa: French national guidelines (PNDS) for diagnosis and treatment]. Ann Dermatol Venereol. 2017 Jan;144(1):6-35. doi: 10.1016/j.annder.2016.07.016. Epub 2016 Dec 5. French. PMID 27931749
- [Background] Lustre A, Levé-Corset I, Leeuwin G, Launay C, Blondy MF, Michaud MT, et al. Soins infirmiers de l'épidermolyse bulleuse. Rev Fr Allergol Immunol Clin. 2001 ; 41(7) : 659-663.
- [Background] Jérôme Palazzolo, Julie Arnaud, Anxiété et performance : de la théorie à la pratique, Annales Médico-psychologiques, revue psychiatrique, Elsevier, Volume 171, Issue 6, July 2013, Pages 382-388.
- [Background] Bandura, A. Auto-efficacité. Le sentiment d'efficacité personnelle (Trad. J. Lecomte). Bruxelles : De Boeck. 2003.
- [Background] Gadbois, C., Aides-soignantes et infirmières de nuit, conditions de travail et vie quotidienne, Paris : Etudes et Recherches, 1981.
- [Background] Van Daele A., Le stress chez les médecins généralistes : une approche transactionnelle, In B. Gangloff (Ed.), satisfactions et souffrances au travail (60-67), Paris : l'Harmattan.
- [Background] Verquerre R., Rusinek-Nisot, Etude du stress chez des infirmiers, In R.Jacob et R. Laflamme (Eds), Stress, santé et intervention au travail, (61-71), Québec : Presses Inter Universitaires.
- [Background] Borteyrou X, Bruchon-Schweitzer M, Spielberger CD. [The French adaptation of the STAXI-2, C.D. Spielberger's State-trait anger expression inventory]. Encephale. 2008 Jun;34(3):249-55. doi: 10.1016/j.encep.2007.06.001. Epub 2007 Oct 10. French. PMID 18558145